CLINICAL TRIAL: NCT04286256
Title: Using Motivational Interviewing To Reduce Parental Risk-Related Behaviors For Early Childhood Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1107M02642
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Caries,Dental; Caries
Keywords: Early Childhood Caries; Motivational Interviewing
MeSH Terms: conditions — Dental Caries | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group received motivational interviewing.
  Interventions: Behavioral: Motivational Interviewing
- Control Group (No Intervention): The control group received standard information only.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Participants/caregivers will receive several telephone-based and in-person motivational interviewing sessions along with specific oral health recommendations.
  Arms: Treatment Group

SUMMARY:
The study's aim was to investigate if a motivational interviewing intervention (MI) improved oral self-care behaviors of AIAN caregivers of infants and determine if the MI intervention promoted positive changes in caregivers' ECC risk-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

- healthy mothers/caregivers of infants

Exclusion Criteria:

* Subjects with recent antibiotic use (within 3 months)
* Subjects on any medication that is immunosuppressive
* Subjects who self-report they have xerostomia due to medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2012-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Concentration of Lactobacilli | Baseline, 8 months
  Oral concentration of Lactobacilli will be measured using a Caries Risk Test (CRT). Outcome will be reported in colony-forming units per milliliter (CFU/mL).
Change in Concentration of Mutans Streptococcus | Baseline, 8 months
  Oral concentration of Mutans streptococcus will be measured using a Caries Risk Test (CRT). Outcome will be reported in colony-forming units per milliliter (CFU/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Blue, BSDH, MS, DHSc, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Blue CM, Arnett MC, Ephrem H, Lunos S, Ruoqiong C, Jones R. Using motivational interviewing to reduce parental risk related behaviors for early childhood caries: a pilot study. BMC Oral Health. 2020 Mar 29;20(1):90. doi: 10.1186/s12903-020-1052-6. PMID 32223762